CLINICAL TRIAL: NCT02313753
Title: Evaluation of the Coping Long Term With Active Suicide Program
Acronym: CLASP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Ivan Miller, Director, Psychosocial Research, Butler Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MH101129
Record Dates: First submitted 2014-12-05; First posted 2014-12-10 (Estimated); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Suicide
MeSH Terms: conditions — Suicide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SAFE (Active Comparator): Safety Assessment and Follow-up Evaluation Protocol
  Interventions: Behavioral: SAFE
- CLASP (Experimental): Coping Long Term with Active Suicide Program Protocol
  Interventions: Behavioral: CLASP

INTERVENTIONS:
Behavioral: CLASP
  Arms: CLASP
Behavioral: SAFE
  Arms: SAFE

SUMMARY:
The purpose of this study is to evaluate the utility of the Coping Long Term with Active Suicide Program (CLASP) for reducing suicidal behavior.

ELIGIBILITY:
Inclusion Criteria:

1. Current patient at Butler Hospital
2. Suicide attempt or suicidal ideation with intent to make a suicide attempt within 48 hours of hospitalization as indicated on the hospital chart and confirmed by administration of the C-SSRS
3. Age > 18 years
4. Have a reliable telephone
5. Ability to speak, read, and understand English well to complete the procedures of the study

Exclusion Criteria:

1. Current psychotic symptoms severe enough to impair study participation
2. Participation in a treatment program with established efficacy in preventing suicidal behavior
3. Cognitive impairment which would interfere with adequate participation in the project (MMSE< 20).

4. Currently in state custody or pending legal action 5. Already enrolled current or previous CLASP trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 224 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
A composite composed of the number of participants with either a suicide attempt or death by suicide | 52 weeks following discharge from hospital
  As assessed by both the Columbia Suicide Severity Rating Scale and record review

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States